CLINICAL TRIAL: NCT06493877
Title: Respiratory Rehabilitation Based on Eccentric Exercice on Treadmill After Thoracic Surgery: a Randomized Clinical Trial
Brief Title: Respiratory Rehabilitation Based on Eccentric Exercice on Treadmill After Thoracic Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Europea de Madrid (Other)
Responsible Party: Principal Investigator, Teresa Fernandez Pardo, Msc, Universidad Europea de Madrid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 082/24
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Thoracic Surgery; Breathing; Muscle
Keywords: "thoracic surgery"; "eccentric training"; "pulmonary rehabilitation"
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aerobic exercice on a treadmill with a negative slope (Experimental): The aerobic exercise will be developed in interval mode, on a treadmill with a negative slope of up to -6% for the intervention group, performing a 2-minute interval with the workload estimated in METS, followed by another 4-minute interval with half the work intensity. It will last between 20 and 30 minutes. The intensity or workload will be individualized (between low and medium), according to the functional status of each participant and will be gradually increased depending on their tolerance. The working heart rate will be between 60% and 80% of the theoretical maximum HR, the oxygen saturation. It should never go below 90% and the subjective perception of effort according to the modified Borg scale will have its objective between 4 and 6 maximum. The treadmill used is the Commercial X22i model from Nordictrack, with a maximum slope of -6º.
  Interventions: Other: Retraining program after thoracic surgery
- Aerobic exercice on a treadmill with a positive slope (Active Comparator): The aerobic exercise will be carried out in interval mode, on a treadmill with a positive slope, performing a 2-minute interval with the workload estimated in METS, followed by another 4-minute interval with half the work intensity. It will last between 20 and 30 minutes. The intensity or workload will be individualized (between low and medium), according to the functional status of each participant and will be gradually increased depending on their tolerance. The working heart rate will be between 60% and 80% of the theoretical maximum HR, the oxygen saturation It should never go below 90% and the subjective perception of effort according to the modified Borg scale will have its objective between 4 and 6 maximum. The treadmill used is the Commercial X22i model from Nordictrack, with a maximum slope of 40º
  Interventions: Other: Retraining program after thoracic surgery
- Aerobic exercice on a cycle ergometer (Active Comparator): The aerobic exercise will be carried out in interval mode, on a cycle ergometer, performing a 2-minute interval with the estimated workload in watts, followed by another 4-minute interval with half the work intensity. It will last between 20 and 30 minutes. The intensity or workload will be individualized (between low and medium), according to the functional status of each patient and will be gradually increased depending on her tolerance. The working heart rate will be between 60% and 80% of the theoretical maximum HR, the oxygen saturation should never drop below 90% and the subjective perception of effort according to the modified Borg scale will have its objective between 4 and 6. maximum.
  Interventions: Other: Retraining program after thoracic surgery

INTERVENTIONS:
Other: Retraining program after thoracic surgery — An effort retraining program will be carried out, with respiratory physiotherapy, muscle strengthening exercises and aerobic exercise, for four weeks, every other day, with a duration of 75 minutes each session. Both the control and experimental groups will receive a common treatment: Muscle strength and aerobic resistance exercises will be performed following the F.I.T.T principle, working the main muscle groups against resistance (between 40% and 60% RM) performing three sets of ten repetitions of each one. It will begin with a warm-up and then a cool down with stretching. We will apply respiratory physiotherapy techniques to promote ventilation and drainage of secretions.
  Next, the aerobic work is carried out according to the assigned group: treadmill with a positive slope (experimental group), treadmill with a negative slope (control 1) or cycle ergometer (group 2).

SUMMARY:
Thoracic surgeries are frequent and pulmonary rehabilitation is essential, since one of the problems that these patients present is dyspnea when performing aerobic exercise, which limits improvement and in some cases causes them to abandon physical exercise. Thanks to carrying out a correct effort retraining program, combining respiratory physiotherapy with therapeutic exercise, patients with respiratory pathologies manage to improve lung capacity and ventilatory mechanics, increase muscle strength and aerobic resistance, prevent long- term complications, reduce fatigue and, ultimately, improve your quality of life.

Likewise, it is important to find the most appropriate type of muscular work that produces more benefits in the short and medium term to optimize our resources.The objective of the study is to demonstrate the effectiveness of eccentric training in patients who have undergone thoracic surgery, in terms of strength, lung capacity, functionality and quality of health in the short and medium term.

For this purpose, a randomized clinical trial has been designed, with a blinded examiner, following the CONSORT guideline for clinical trials and the ethical principles of the Declaration of Helsinki. A total sample of 57 subjects has been estimated. The study is aimed at patients after scheduled thoracic surgery. A program of 12 group sessions spread over 4 weeks will be carried out. Each of them will last 75 minutes and will include strength and respiratory physiotherapy exercises, common to all subjects.

Aerobic interval training will depend on the group assigned: treadmill with negative slope (experimental group), treadmill with positive slope (control group 1) or cycle ergometer (control group 2). On the first and last day of treatment, as well as one month after completing the intervention, the following variables will be measured: thickness, cross-sectional area and ultrasound intensity of the rectus femoris; diaphragmatic excursion and thickness; 6 minute walk test; Borg scale; maximum respiratory pressures; sit-to-stand test; grip strength in both hands; spirometric assessment of FEV1 and SF-12 health quality questionnaire. a

ELIGIBILITY:
Inclusion Criteria:

* Subjects >18 years.
* Thoracic surgery in the previous 75 days
* Present dyspnea grade 2 - 3 on the mMRC scale.
* Cognitive and functional level sufficient to understand, learn and carry out the exercise program.
* Not have contraindications to perform physical training.
* Active collaborators.

Exclusion Criteria:

* Severe intolerance to exertion due to untreated cardiac arrhythmias, ischemia during low intensity exercise (anginas unstable), severe pulmonary hypertension, heart failure (NYHA III or IV)
* Pulmonary embolism with anticoagulant treatment less than 5 days.
* Recent cardiovascular events such as congestive heart failure, angioplasties or cardiac surgeries of less than four weeks' duration, valvular alterations requiring surgical correction, myopericarditis, ventricular arrhythmias caused by exercise.
* Kidney failure requiring dialysis.
* Patients with uncontrolled bronchospasm due to intrinsic asthma.
* Patients undergoing post-surgery chemotherapy treatment.
* Adverse effects that occurred during the development of the treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Rectus femoral thickness | Baseline, 3 weeks, 2 months
  The dominant quadriceps (defined by the leg that is usually used to climb stairs or kick a ball) is measured, with the patient's starting position being supine with the knee completely extended and relaxed. While previous studies suggested a minimum of 30 minutes of rest before performing the ultrasound, more recent studies indicate that 5 minutes after adopting the supine position, measurements normalize. There is no consensus on the measurement point, but it is proposed to place the probe at the midpoint of the muscle length (50% rule), taking the greater trochanter and proximal edge of the patella as reference. It is also advisable to place the probe midway between the medial and lateral edges of the muscle. Once the placement point of the probe has been determined, it is placed as perpendicular as possible to the skin using a generous amount of transducer gel and exerting the minimum possible pressure to avoid compression of the dermal surface and muscle distortion.
Diaphragmatic excursion | Baseline, 3 weeks, 2 months
  A convex probe of 2.5 to 3.5 MHz is used. In obese subjects, to have better visibility, the frequency chosen is 1.5 MHz.
  The subjects are in a supine position, with the head of the stretcher flat and their legs bent at 30-45º. The probe is positioned firmly below the right costal arch and on the line drawn corresponding to the middle of the clavicle, orienting it cranially. At that point, the dome of the right hemidiaphragm is visualized, appearing as a thick hyperechoic line. The highest diaphragmatic position is sought, which is the part of the diaphragm that produces the most craniocaudal excursion, and the transducer is kept firmly in position during the phases of the respiratory cycle and measurements of tidal volume breathing. The M mode modality is then activated, which provides us with the diaphragmatic movement pattern, placing the M beam line around 30º in the posterior part of the cranio-caudal midline: cranio-caudal diaphragmatic excursions.
Diaphragm thickness | Baseline, 3 weeks, 2 months
  The measurement of the thickness of the diaphragm is taken in the right hemidiaphragm since it is more accessible than the left through its hepatic window. To evaluate the thickness, a linear probe at 10-12MHz is used, placing it perpendicular to the intercostal space between the 9th and 10th rib, in the anterior part of the axillary line. At this level, 3 parallel layers with different echogenicity are observed corresponding to the pleura, the diaphragm and the peritoneum. The measurement is carried out with M mode, where the image is frozen in an unforced expiration (representing the functional residual capacity) and in a maximum inspiration. The distance between the inner edge of the pleural line and the inner edge of the peritoneal line is measured. The measurement is carried out three times and the average of the three is taken.
6MWT | Baseline, 3 weeks, 2 months
  In this test, the patient is asked to walk the maximum possible distance along a minimally traveled 30-meter corridor for a period of 6 minutes following a standardized protocol. The primary outcome will be the distance walked in 6 minutes measured in meters, with several reference equations that allow normality values to be calculated. It is essential to follow a standardized 6MWT methodology to obtain reproducible and reliable results, which is why the indications of the SEPAR Manual of Procedures are followed.
Perceived effort | Baseline, 3 weeks, 2 months
  It is measured through the Borg scale, which consists of a vertical scale from 0-10 that relates the perceived effort when making physical effort with a numerical value that ranges from 0 (minimal effort) to 10 (extreme effort).
Measurement of maximum respiratory pressures (MIP and PEM). | Baseline, 3 weeks, 2 months
  The pressure gauge we use is the RP Check. To measure PEM, the patient must insert the mouthpiece into his or her mouth, with the bite blocks between the teeth; You should inhale as much air as possible until you completely fill your lungs (to full lung capacity) and then exhale as hard as possible and for as long as possible (1.5 seconds minimum). To measure PIM, the patient must insert the mouthpiece into his mouth, exhale as much air as possible to empty his lungs until reaching the residual volume, and then inhale with as much effort as possible and for as long as possible (minimum 1.5 seconds). We perform three consecutive measurements of each one, allowing the patient to rest one minute between each one, and we note the best result.
Functional capacity | Baseline, 3 weeks, 2 months
  Through the 30-second sit to stand test. We previously measured basal oxygen saturation and heart rate; The patient performs the test with his arms crossed over his chest; We time 30 seconds and write down the result. Next, we measure the saturation of oxygen and heart rate.
Grip strength measurement in both hands | Baseline, 3 weeks, 2 months
  With the Hand Grip Dynamometer Kern Map Version 1.2 dynamometer, taking into account the dominant hand and possible injuries to the upper limbs that may interfere with the test result.
Spirometric assessment of FEV1 | Baseline, 3 weeks, 2 months
  We performed three consecutive measurements with the Vitalograph copd-6™. You need to enter your age, height and gender. The patient must inhale completely, hold the breath, gently bite the mouthpiece and then blow as hard as they can for 6 seconds, allowing them to rest for a minute between each one and we will record the best result.
Life quality | Baseline, 3 weeks, 2 months
  SF-12 Health Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Fernandez Pardo, Msc, Study Director — Universidad Europea de Madrid
Locations (1):
- Hospital Universitario Ramon y Cajal, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No